CLINICAL TRIAL: NCT05526898
Title: Multi-Center, Randomized Controlled Trial Evaluating the Effect of Adipose Tissue Processed With the SyntrFuge™ System for Knee Osteoarthritis
Brief Title: Evaluating the Effect of Adipose Tissue Processed With the SyntrFuge™ System for Knee Osteoarthritis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Syntr Health Technologies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SHT-SYN-03
Record Dates: First submitted 2022-08-31; First posted 2022-09-02 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Knee Osteoarthritis
Keywords: Microsized Fat Tissue; Adipose Tissue; Fat Transfer; Knee Osteoarthritis; Orthopedic Surgery
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Triamcinolone

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- SyntrFuge System (Experimental): Adipose tissue microsized via the SyntrFuge System
  Interventions: Device: SyntrFuge System
- Standard of Care (Other): Steroid Injection
  Interventions: Drug: Triamcinolone Injection

INTERVENTIONS:
Device: SyntrFuge System — Microsized Adipose Tissue
  Arms: SyntrFuge System
Drug: Triamcinolone Injection — Corticosteroid
  Arms: Standard of Care

SUMMARY:
This is an multi-center study with the aim of evaluating the efficacy of adipose tissue processed with the SyntrFuge™ system in Orthopedic Surgery, specifically Knee Osteoarthritis. Patients will be enrolled to the treatment group with adipose tissue processed with the SyntrFuge™ system followed by an injection of autologous microsized adipose tissue in the treatment sites or Standard of Care.

ELIGIBILITY:
Inclusion Criteria

* Subjects aged of 35-80 years old
* Patients with knee osteoarthritis grade II, III, and IV Kellgren-Lawrence
* Chronic knee pain or symptoms for at least 3 months
* BMI between 20 and 34.9
* Willing and able to read and sign the informed consent and other study materials
* Written informed consent has been obtained prior to any study-related procedures
* Written Authorization for Use and Release of Health and Research Study Information has been signed
* Subjects are ambulatory
* Subject is willing and able to comply with study instructions and commit to all follow-up visits for the duration of the study
* Females of childbearing potential must have a negative urine pregnancy test result and not be lactating
* Subject is in good general health and free of any systemic disease state or physical condition that might impair evaluation or which in the Investigator's opinion, exposes the Subject to an unacceptable risk by study participation

Exclusion Criteria:

* Subjects with previous traumatic lesion (tibial fracture, osteothomy) of the knee
* Subjects with osteonecrosis
* Subjects with meniscal surgery in the previous 6 weeks
* Subjects with gout, hyperlipidemia
* Subjects without decisional capacity
* Subjects with inflammatory arthritis
* Subjects with active infection
* Subjects with any uncontrolled systemic disease
* Subjects with a history of severe allergic/anaphylactic reactions or multiple allergies
* Subjects planning to become pregnant, are pregnant, or are breast-feeding
* Subjects with history or current evidence of drug or alcohol abuse within 36 months prior to screening visit
* Subjects who have active autoimmune disease
* Subjects who have coagulation disorders
* Subjects who have received any other therapy, which, in the opinion of the investigator, could interfere with safety or efficacy evaluations
* Subjects with current enrollment in an investigational drug or device study or participation in such a study within 30 days of entry into this study
* Subjects with any other condition that, in the opinion of the investigator, makes the subject inappropriate to take part in this study
* Subjects who have received anti-coagulation, anti-platelet, or thrombolytic medications (e.g., warfarin), anti- inflammatory drugs (NSAIDs, e.g., aspirin, ibuprofen), or other substances known to increase coagulation time from 7 days pre- to 3 days post injection. A wash out period of 7 days is allowed
* Subjects who have undergone immunosuppressive therapy, chemotherapy, biologics or systemic corticosteroids within 3 months prior to each study visit.
* No intra-articular injection of corticosteroids within the last 24 weeks
* No intra-articular injection of any other cellular therapy within the last 24 weeks

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 176 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
WOMAC | 6 months, 12 months, 24 months
  Change of WOMAC Score from Baseline

SECONDARY OUTCOMES:
Knee Injury and Osteoarthritis Outcomes Score (KOOS) | 6 months, 12 months, 24 months
  Change in Knee Injury and Osteoarthritis Outcomes Score (KOOS) Over Time
Single Assessment Numerical Evaluation | 6 months, 12 months, 24 months
  Change in Single Assessment Numerical Evaluation (SANE) Over Time

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Irvine Site 1, Irvine, California
  - Irvine Site 2, Irvine, California

IPD SHARING:
Plan to Share IPD: No